CLINICAL TRIAL: NCT01085994
Title: Procalcitonin-guided Algorithms of Antibiotic Stewardship in the Intensive Care Unit: Systematic Review and Meta-analysis
Brief Title: Procalcitonin Monitoring May Decrease Antibiotic Use in the Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Athens (Other)
Responsible Party: Petros Kopterides, MD, University of Athens Medical School, 2nd Critical Care Department, "Attiko" University Hospital
Other Study IDs: PCT-2010
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-01

CONDITIONS: Sepsis
Keywords: antibiotics; resistance; bio-marker; procalcitonin; algorithm; critically ill
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Procalcitonin-guided group
  Interventions: Other: Literature search
- Routine practice group
  Interventions: Other: Literature search

INTERVENTIONS:
Other: Literature search — Literature search followed by systematic review and meta-analysis

SUMMARY:
Sepsis is common and is associated with significant mortality, morbidity and health-care costs. Unfortunately, its diagnosis is not straightforward because its signs and symptoms are neither specific nor sensitive; in addition, microbiological cultures lack specificity, sensitivity and are plagued by high turn-around times. Because the delay in the institution of antimicrobial therapy may be deleterious, broad-spectrum antibiotics are widely used in ICU-patients, even when they are not needed. Procalcitonin may not be the long sought for bio-marker to establish the diagnosis of sepsis but may help decrease the duration of the administered antibiotic courses once they are started.

DETAILED DESCRIPTION:
Recently, a number of studies have shown the utility of procalcitonin (PCT) measurements in reducing the duration of antibiotic treatment in patients with respiratory tract infections presenting to the primary care setting or the emergency department. However, it remains unclear if a similar strategy can be effectively and safely implemented in the critical care setting. We attempt to address the controversy on this issue, by collecting, analyzing and interpreting the currently available relevant evidence. To this end, a systematic review and meta-analysis of the randomized controlled trials reporting on the outcomes of critically ill septic patients managed with or without a procalcitonin-based algorithm will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled trials (RCTs) that report on the outcomes of critically ill patients managed with a procalcitonin-guided algorithm versus routine practice.
* Participants of any age with proven or suspected sepsis will be considered. - As routine practice, the investigators will consider the institution and discontinuation of antibiotics by the attending physicians with the aid of clinical signs, symptoms, microbiological data, well established laboratory parameters (i.e., white blood cell count) and widely accepted guidelines but without the knowledge of PCT values. The investigators will set no limitations regarding the time, country or language of publications. The investigators will search for trials conducted in critically ill neonates and children.

Exclusion Criteria:

* The investigators will exclude studies that are not RCTs and studies performed outside the ICU, namely in the primary care setting, the emergency department or the clinic.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will systematically search PubMed, Scopus and the Cochrane Central Register of Controlled Trials to identify relevant randomized controlled trials by using the following search terms: procalcitonin AND ("critically ill" OR "intensive care" OR "critical care"). The reference lists of the initially retrieved articles will also be reviewed. Abstracts of conference proceedings will not be sought because they commonly present data that differ from the full publications. Finally, the corresponding authors of each one of the included studies will be contacted by e-mail for additional information and clarifications if needed.
Sampling Method: Probability Sample
Dates: Start 2010-01; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Duration of antibiotic treatment for the first episode of infection
Total duration of antibiotic therapy
Antibiotic-free days at 28 days after study enrollment

SECONDARY OUTCOMES:
28-day mortality
In-hospital mortality
Length of ICU stay
Length of hospital stay
Days free of mechanical ventilation at 28 days after study enrollment
Rates of relapsed/persistent infection
Rate of superinfection
Financial cost of implementing a procalcitonin-based algorithm: purchase of the laboratory equipment/reagents, cost of the administered antibiotics, charges for hospital stay etc

CONTACTS AND LOCATIONS:
Overall Officials: Petros Kopterides, MD, Principal Investigator — University of Athens Medical School
Locations (1):
- University of Athens - Medical School, Athens, Greece

REFERENCES:
- [Background] Schuetz P, Christ-Crain M, Thomann R, Falconnier C, Wolbers M, Widmer I, Neidert S, Fricker T, Blum C, Schild U, Regez K, Schoenenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Mueller B; ProHOSP Study Group. Effect of procalcitonin-based guidelines vs standard guidelines on antibiotic use in lower respiratory tract infections: the ProHOSP randomized controlled trial. JAMA. 2009 Sep 9;302(10):1059-66. doi: 10.1001/jama.2009.1297. PMID 19738090
- [Background] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Background] Moher D, Liberati A, Tetzlaff J, Altman DG; PRISMA Group. Preferred reporting items for systematic reviews and meta-analyses: the PRISMA statement. Ann Intern Med. 2009 Aug 18;151(4):264-9, W64. doi: 10.7326/0003-4819-151-4-200908180-00135. Epub 2009 Jul 20. No abstract available. PMID 19622511
- [Result] Kopterides P, Siempos II, Tsangaris I, Tsantes A, Armaganidis A. Procalcitonin-guided algorithms of antibiotic therapy in the intensive care unit: a systematic review and meta-analysis of randomized controlled trials. Crit Care Med. 2010 Nov;38(11):2229-41. doi: 10.1097/CCM.0b013e3181f17bf9. PMID 20729729